CLINICAL TRIAL: NCT03308149
Title: Predictability of the Effects of Facet Joint Infiltration in the Degenerate Lumbar Spine When Assessing MRI Scans
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ulf Krister Hofmann, Principal Investigator, University Hospital Tuebingen
Other Study IDs: 503/2016BO2
Record Dates: First submitted 2017-09-28; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Infiltration Facet Joint
MeSH Terms: interventions — Triamcinolone; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: infiltration with triamcinolone and bupivacaine — facet joint infiltration

SUMMARY:
Fifty MRI scans of patients with chronic lumbar back pain were graded radiologically using a wide range of classification and measurement systems. The reported effect of facet joint injections at the site was recorded and a comparative analysis performed.

ELIGIBILITY:
Inclusion Criteria:

* patients who had received inpatient gradual diagnostics for chronic lumbar back pain
* monosegmental facet joint infiltration on the first day of inpatient gradual diagnostics
* clearly stated pain relief in percentage (%) for that specific infiltration in the medical documentation
* pain level prior to infiltration needed to be clearly documented
* a high-quality MRI available before infiltration.

Exclusion Criteria:

* ositive history of lumbar surgery or the presence of artificial implants in the area of interest

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who had received inpatient gradual diagnostics in our department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Correlation of radiologic findings and reported pain relief | Improvement in pain level within 24 hours
  Pain relief is assessed as an improvement in % on the NRS. Radiologic findings consist of numerous classification systems and measurement techniques to evaluate and classify spinals and neural foramen stenosis, like for example as suggested by Schizas, or the sagittal diameter of the spinal canal

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Hofmann, M.D., Principal Investigator — Department of Orthpaedic Surgery, University Hospital of Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Orthopaedics, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
General data file from which statistical analyses were performed may be requested from the authors after publication

REFERENCES:
- [Derived] Hofmann UK, Keller RL, Walter C, Mittag F. Predictability of the effects of facet joint infiltration in the degenerate lumbar spine when assessing MRI scans. J Orthop Surg Res. 2017 Nov 21;12(1):180. doi: 10.1186/s13018-017-0685-x. PMID 29162138